CLINICAL TRIAL: NCT04303819
Title: The Effect of Exenatide on Fasting Bile Acids in Newly Diagnosed Type 2 Diabetes Mellitus Patients, a Pilot Study
Brief Title: The Effect of Exenatide on Fasting Bile Acids
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Lihong Liu, professor, Beijing Chao Yang Hospital
Other Study IDs: 20131212
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes Mellitus in Obese
MeSH Terms: interventions — Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly diagnosed T2DM participants: newly diagnosed T2DM participants without anti-diabetic drugs intake
  Interventions: Drug: Exenatide treatment

INTERVENTIONS:
Drug: Exenatide treatment — 12 weeks of exenatide injection, 5 μg twice a day by subcutaneous injection for 4 weeks, followed by 10 μg twice a day for 8 weeks, as recommended by the drug manufacturer.
  Other Names: exenatide

SUMMARY:
Newly diagnosed T2DM participants without hypoglycemic drugs intake were retrospective analyzed. Plasma total bile acids in fasting state (FTBAs) and other parameters were compared before and after exenatide treatment and correlation analysis between changes of FTBAs and glycemic parameters.

DETAILED DESCRIPTION:
Newly diagnosed T2DM participants without hypoglycemic drugs intake were retrospective analyzed. Plasma total bile acids in fasting state (FTBAs) and other parameters were tested at baseline. Then exenatide were applied to the T2DM participants for 12 weeks. FTBAs and glycemic parameters were measured again after exenatide treatment, and correlation analysis between changes of FTBAs and glycemic parameters were conducted to investigate the role of BAs in the glycemic control effect of exenatide.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed T2DM patients

Exclusion Criteria:

* History of hepatobiliary or pancreatic diseases
* History of anti-diabetic drugs intake
* Change of anti-dyslipidemia therapy regimen
* Estimated glomerular filtration rate less than 60 mL/min/1.73 m^2
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma total bile acids in fasting state | 12 weeks
  reported in μmol/L

SECONDARY OUTCOMES:
fasting plasma glucose | 12 weeks
  reported in mmol/L
Glycated hemoglobin A1c | 12 weeks
  reported in %
C-peptide | 12 weeks
  reported in mU/L
Fasting serum insulin | 12 weeks
  reported in mU/L
Body mess index | 12 weeks
  reported in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Boyu Li, PHD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-yang hospital, Beijing, China

REFERENCES:
- [Derived] Li B, Hu Y, Wang G, Liu L. The effect of exenatide on fasting bile acids in newly diagnosed type 2 diabetes mellitus patients, a pilot study. BMC Pharmacol Toxicol. 2020 Jun 15;21(1):44. doi: 10.1186/s40360-020-00422-5. PMID 32539783